CLINICAL TRIAL: NCT05305456
Title: A Randomized, Double-blind, Placebo-controlled, Multicenter Clinical Trial of Tanreqing Capsule Efficacy and Safety in the Treatment of COVID-19 (Mild and Common Type)
Brief Title: Clinical Trial Scheme of Tanreqing Capsules in the Treatment of COVID-19
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Jiangsu Famous Medical Technology Co., Ltd. (Industry)
Collaborators: Ruijin Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: FM-P8-2022032501
Record Dates: First submitted 2022-03-30; First posted 2022-03-31 (Actual); Last update posted 2022-12-06 (Actual); Status verified 2022-11

CONDITIONS: Novel Coronavirus Pneumonia
Keywords: mild, common
MeSH Terms: conditions — Lymphoma, Follicular | interventions — tanreqing

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tanreqing capsule (Experimental): 3 capsules per time, 3 times a day，7 days of treatment
  Interventions: Drug: Tanreqing capsule
- Tanreqing capsule simulator (Placebo Comparator): 3 capsules per time, 3 times a day，7 days of treatment
  Interventions: Drug: Tanreqing capsule simulator

INTERVENTIONS:
Drug: Tanreqing capsule — 3 capsules per time, 3 times a day
  Other Names: Basic treatment: Vitamin C effervescent tablet, 1g, once a day, warm boiled water after brewing, continuous administration for 7 days.
  Arms: Tanreqing capsule
Drug: Tanreqing capsule simulator — 3 capsules per time, 3 times a day
  Other Names: Basic treatment: Vitamin C effervescent tablet, 1g, once a day, warm boiled water after brewing, continuous administration for 7 days.
  Arms: Tanreqing capsule simulator

SUMMARY:
This study was conducted in a randomized, double-blind, placebo-controlled, multicenter clinical trial design. Two groups were designed, the experimental group and the placebo control group. Patients in both groups received basic treatment with vitamin C effervescent tablets. Tanreqing capsule was added to basic treatment in the experimental group, and placebo was added to basic treatment in the control group. The treatment course was 7 days, and the observation period was set to 7 days, with a daily visit.

DETAILED DESCRIPTION:
The purpose of this study was to evaluate the efficacy and safety of Tanreqing capsule in the treatment of mild and common COVID-19. The trial was a randomized, double-blind, placebo-controlled, multicenter clinical trial design. A total of 480 patients were divided into 2 groups: experimental group and control group 3:1. Patients in both groups received basic treatment with vitamin C effervescent tablets. Tanreqing capsule was added to basic treatment in the experimental group, and placebo was added to basic treatment in the control group. The treatment course was 7 days, and the observation period was set to 7 days, with a daily visit.

ELIGIBILITY:
Inclusion Criteria:

1. According to the Diagnosis and Treatment Plan for Pneumonia Infected by novel coronavirus (Trial Version 9), those who are in line with the diagnosis of novel coronavirus pneumonia and whose clinical classification is light and ordinary；
2. Aged greater than 18, with no gender limitation;
3. Symptom score greater than or equal 3 points;
4. Voluntarily accept the drug treatment and sign the informed consent.

Exclusion Criteria:

1. Patients with severe primary respiratory diseases or other pathogenic microbial pneumonia that needs to be differentiated from COVID-19;
2. immune deficiency disease, or use of immunosuppressants or glucocorticoids in the last 3 months;
3. pregnant and lactating women;
4. People with allergic constitution (allergic to more than two drugs or food or known allergic to the drug used in this study);
5. mentally ill persons or persons without self-awareness;
6. Patients whose expected survival time from screening is not more than 48 hours; (7) those who have been intubated or mechanically ventilated at the time of screening;

(8) In patients with serious primary diseases of heart, brain, liver and kidney, ALT and AST were 1.5 times higher than the upper limit of normal value; (9) Other conditions that the investigator considers inappropriate for clinical trial participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 480 (Actual)
Dates: Start 2022-03-28 (Actual); Primary Completion 2022-06-02 (Actual); Study Completion 2022-08-31 (Actual)

PRIMARY OUTCOMES:
The time from the first dose to sustained clinical recovery | 8 days
  Symptom domains and minors disappear completely within 7 days treatment period after randomization, and maintain it for 2 days without recurrence and the disease don't aggravate

SECONDARY OUTCOMES:
Novel coronavirus N and ORF gene changes | 8 days
  Nucleic acid detection was performed on the 0, 1, 2, 3, 4, 5, 6 and 7 days respectively.
  The fluorescent quantitative PCR method was used to determine the Ct value of N gene and ORF gene in novel coronavirus nucleic acid detection. Negative: no Ct value or Ct value>40. Positive: Ct value<35. Ct value (cycle threshold) refers to the Ct value of nucleic acid detection, that is, the number of cycles required when the pcr fluorescence signal reaches the threshold.
The time from the first dose/first testing positive of virus to testing sustained negative of virus within 7 days treatment period after randomization | 8 days
  Testing sustained negative of virus was defined two consecutive (at least 24 hours apart) nasal swabs with new coronavirus nucleic acid detection CT values 35 ,and the negative event date was defined by first negative occurrence.
Effective rate of wind heat attacking lung syndrome | 8 days
  The time from the first dose to sustained clinical improvement defined total scores for symptom domains and minors was <3 within 7 days treatment period after randomization.
Duration of disappearance of main symptoms of wind heat attacking lung syndrome | 8 days
  The time from the first dose to sustained complete disappearance within 7 days treatment period after randomization for every symptom domain, and these two outcomes definition were similar to the primary outcome.
Weight conversion rate (ratio of light type to ordinary type and ordinary type to heavy type) | 90 days
  Proportion of patient experiencing progression to severe illness diagnosed by Trial draft version 9 of Diagnosis and Treatment Protocol for novel Coronavirus pneumonia within 7 days treatment period after randomization, during period from the end of 7 days treatment period to discharged from hospital and 3-month follow-up period after discharge.

CONTACTS AND LOCATIONS:
Overall Officials: Zhao Ren, PhD, Principal Investigator — Ruijin Hospital affiliated to Shanghai Jiaotong University School of Medicine (North Hospital)
Locations (2):
- China (2):
  - Huashan Hospital Affiliated to Fudan University, Shanghai, Shanghai Municipality
  - Shanghai Public Health Clinical Center, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: Undecided